# 初治成人急性髓系白血病患者中标准 "3+7"方案与维奈克拉联合 CACAG 方案的多 中心前瞻随机对照研究

## 研究方案

版本号: v1.0, 版本日期: 2024年3月11日

一、 研究背景、国内外研究现状及最新进展、突出临床问题与科学问题, 并附主要参考文献目录

#### 1. 研究背景

20世纪70年代起,DA或IA方案(3+7方案)成为了AML的标准诱导治疗方案,在年轻成人AML患者中完全缓解率达到60-70%<sup>[1,2]</sup>。近40年研究中发现通过增强化疗药物剂量、增加化疗药物种类或联合其他靶向药物,可以提高部分携带特定分子学异常的AML患者的治疗反应率,但成人AML总体预后并无明显改善。且AML多种化疗药物耐药的机制存在共同性,如蒽环类药物、嘧啶类抗代谢药物阿糖胞苷等存在共同的耐药机制<sup>[3]</sup>。而且白血病细胞一旦对一种药物产生耐药,往往多种药物皆存在耐药情况<sup>[4]</sup>。

AML的治疗决策在近几十年主要围绕着化疗方案的强度和不同化疗药物的组合,缺少突破性进展。虽然国内外不断有治疗AML的新药上市,包括靶向BCL-2(B-cell lymphoma-2,B淋巴细胞瘤-2)的维奈克拉,靶向FLT3(Fms-like tyrosine kinase, FMS样的酪氨酸激酶3)的米哚妥林和吉瑞替尼,靶向IDH1(i socitrate dehydrogenase soluble 1,可溶性异柠檬酸脱氢酶1)、IDH2的艾伏尼布和恩西地平,针对CD33的GO以及柔红霉素和阿糖胞苷的脂质体复合物CPX-

351<sup>[5]</sup>及IDH2抑制剂等。新药在临床取得了一定的效果<sup>[5-9]</sup>,改善了部分携带特定分子学异常、老年患者及不能耐受强化疗患者的治疗效果,但均替代不了蒽环类药物的重要地位,且初诊的成人AML患者总体预后并无明显改善,仍有约30%的患者因诱导失败或疾病复发而成为复发难治急性白血病<sup>[10]</sup>。

因此,克服原发或复发后的耐药,寻找新的治疗方案提高急性髓系白血病患者诱导化疗的缓解率、提高该类患者治疗疗效、改善患者预后生存有重大的研究价值。

#### 2. 国内外研究现状

#### (1) 蒽环类药物发挥作用的新机制

既往研究认为,蒽环类药物的主要作用机制是通过抑制拓扑异构酶II导致 DNA双链断裂,使细胞启动损伤修复机制,如果未修复成功,细胞则进入凋亡模式。而快速增殖的细胞,例如肿瘤细胞,对DNA损伤更为敏感,这也是化疗药物治疗肿瘤的基本原理之一[11-13]。近年来研究证明,蒽环类药物存在表观遗传调控新机制:

### 1) 既往研究发现以柔红霉素、去甲氧柔红霉素、阿克拉霉素为代表的蒽环 类药物存在新的杀伤白血病细胞的诱导组蛋白释放的表观遗传新机制:

①最近研究证实,柔红霉素、去甲氧柔红霉素、阿克拉霉素为代表的蒽环类药物插入到DNA中时,其糖基部分可以嵌入到DNA双链的沟槽中,并与组蛋白竞争空间,导致核小体崩解组蛋白释放(主要涉及到H3和H4),这些释放的组蛋白随后被其他不同的表观遗传修饰的新生组蛋白所取代<sup>[14-19]</sup>。

②蔥环类药物介导的组蛋白释放影响DNA损伤修复,对于蔥环类药物杀伤白血病细胞作用至关重要。蔥环类药物(除阿克拉霉素外)可以导致DNA双链断裂,DNA双链断裂的早期反应是组蛋白H2AX被磷酸化,是DNA损伤传导信号的首要因素。H2AX的PAGFP修饰(photoactivatable GFP光活化绿色荧光蛋白修饰)并不影响DNA双链断裂后H2AX的磷酸化。申请人团队应用共聚焦显微镜观察柔红霉素处理2h后组蛋白的反应,结果发现柔红霉素可以释放PAGFP-H2AX,暴露于柔红霉素处理后细胞中内源性 γ -H2AX的形成明显弱于依托泊苷处理后,用SDS-PAGE(sodium dodecyl sulfate-polyacrylamide gel electrophoresis,十二烷基硫酸钠-聚丙烯酰胺凝胶电泳)和蛋白免疫印迹(Western blot)分析,经过柔红霉素处理的细胞中 γ -H2AX的产生明显少于依托泊苷处理后的细胞。说明柔红霉素可以

释放组蛋白H2AX,减弱DNA损伤修复反应信号。总而言之,Topo II抑制剂柔红霉素和依托泊苷都会导致DNA双链断裂,但DNA损伤修复反应存在差异(见工作基础部分Figure 6)。证明柔红霉素诱导组蛋白释放,减缓DNA损伤修复信号传导,从而阻碍正常的DNA损伤修复。

- ③蒽环类药物诱导的组蛋白释放对不同细胞系独特的表观遗传染色质状态有选择性,不同蒽环类药物处理后细胞的组蛋白释放情况存在差异,不同的基因组组蛋白释放特征可能与细胞对蒽环类药物的反应存在联系,蒽环类药物诱导的组蛋白释放与局部染色质结构的特征密切相关。用柔红霉素、阿克拉霉素、依托泊苷处理了K562和SU-DHL-4细胞系发现,蒽环类药物在特定染色质特征区域释放组蛋白:阿霉素在有组蛋白H3的36位赖氨酸位点的三甲基化修饰(H3K36me3)的染色质区域释放组蛋白<sup>[18,20]</sup>,柔红霉素及去甲氧柔红与阿霉素效果类似。而阿克拉霉素还会在有组蛋白H3的27位赖氨酸位点的三甲基化修饰(H3K27me3)的染色体区域释放组蛋白。
- ④蔥环类药物组蛋白释放特征不依赖于拓扑异构酶II的抑制、DNA双链断裂或者细胞凋亡。从该角度来说蔥环类药物是一类针对不同表观遗传基因组的选择性调控表观遗传药物。蔥环类药物诱导组蛋白释放后,该区域的染色质随后被新的,有表观遗传修饰的组蛋白所替代,改变了特定区域的表观遗传学修饰。
- 2) <u>申请人既往研究发现阿霉素和柔红霉素(蒽环类药物一种)耐药的急性</u> 髓系白血病细胞中,组蛋白去乙酰化酶HDAC3-AKT-P21-CDK2通路激活,组蛋白 去乙酰化酶抑制剂可以逆转蒽环类药物的耐药,组蛋白修饰状态改变是阿霉素耐 药的重要机制

申请人团队一项研究证明组蛋白的乙酰化修饰与蒽环类药物阿霉素和柔红霉素的耐药密切相关(见工作基础部分Figure 10,11),对蒽环类耐药白血病细胞系和蒽环类敏感细胞系转录组测序发现蒽环类耐药白血病细胞系中组蛋白去乙酰化酶HDAC3显著高表达,组蛋白乙酰化水平降低,HDAC3-AKT-P21-CDK2通路激活,并通过实时荧光定量聚合酶链式反应(qPCR)和Western blot在mRNA和蛋白水平得到验证(见工作基础部分Figure 11)。随后通过HDAC1、2、3及10小分子抑制剂西达本胺(chidamide)抑制HDAC3,发现耐药细胞系增殖能力受到抑制、凋亡增加、细胞周期明显阻滞,并且HDAC3-AKT-P21-CDK2通路在mRNA和蛋白水平明显下调。蒽环类药物耐药白血病细胞中特异性敲除HDAC3后得到相同的结果。西达本胺处理的蒽环类耐药白血病细胞中,上调HDAC3后,可以明显解除西达本胺对于细胞增殖能力的抑制和诱导细胞凋亡的效果,并且HDAC3-AKT-P21-CDK2通

路表达水平恢复。通过机制研究发现,HDAC3蛋白通过结合蛋白激酶(AKT)蛋白,引起AKT去乙酰化,促进AKT磷酸化,磷酸化的AKT进一步增强HDAC3表达,同时HDAC3导致组蛋白乙酰化水平改变,是急性髓系白血病细胞蒽环类药物耐药的重要机制。上述成果已发表于2020年Journal of Experimental & Clinical Cancer Research(影响因子11.16)。进一步研究发现,柔红霉素耐药的急性白血病细胞中,拓扑异构酶II处于低表达状态,但阿克拉霉素仍然可以诱导阿霉素耐药白血病细胞的增殖与凋亡,使其增殖抑制,凋亡增加(结果已完成)。上述结果提示,急性髓系白血病中组蛋白去乙酰化酶抑制剂具有克服蒽环类药物耐药的潜力,组蛋白乙酰化修饰是蒽环类耐药的关键因素,值得在临床上探索。

总的来说,蒽环类药物或许通过改变急性白血病患者的表观遗传学修饰特征治疗白血病,那么直接应用表观修饰药物是否有可能更大的提高患者疗效呢?因此我们提出了双表观药物应用于急性髓系白血病患者诱导化疗的新思路。

#### (2) 表观调控治疗与白血病

白血病的发生发展是一个多阶段、多步骤的过程,随着对急性白血病发病机制研究的不断深入,人们逐渐认识到基因表达改变及调控异常是急性白血病发生的重要机制及预后因素<sup>[5]</sup>,而除遗传学异常外,表观遗传学异常在白血病的发生发展中起着重要的促进和协同作用<sup>[21]</sup>,急性白血病相关基因的表观遗传学改变是当前该领域研究的热点。表观遗传学(Epigenetics)是指在DNA序列不发生改变的情况下,通过表观遗传学修饰如DNA甲基化,RNA甲基化,非编码RNA,组蛋白修饰等影响基因转录及转录后活性,从而调控基因的表达<sup>[20,22-26]</sup>。许多重要的抑癌基因由于其启动子区发生异常DNA甲基化或组蛋白去乙酰化而导致基因表达受到抑制,从而参与白血病发生发展。表观遗传异常具有广泛的影响,和特定的抑癌基因突变相比可以同时影响更多的通路。通常来说,表观遗传过程的异常不是孤立发生的,而是在多个表观遗传调控下进行,最终导致疾病的发生发展。

去甲基化药物目前在急性髓系白血病及骨髓增生异常综合征治疗中应用广泛。 去甲基化药物主要通过与DNA甲基转移酶共价结合,降低该酶转移甲基的生物活 性,从而形成低甲基化的子链,实现去甲基化,达到治疗肿瘤的目的。目前去甲 基化药物主要有地西他滨和阿扎胞苷。但去甲基化药物单药治疗在急性髓系白血 病中疗效并不理想,缓解率仅有15.7-38%<sup>[26,27]</sup>。申请人单位在既往研究中采用地 西他滨与预激方案CAG方案联合组成的DCAG方案,在急性髓系白血病中取得了较 好的疗效<sup>[8,9]</sup>。CAG方案包括重组人粒细胞刺激因子(G-CSF)、阿克拉霉素(A- cla)、阿糖胞苷(Ara-C),其方案在复发、难治急性髓系白血病及骨髓增生异常综合症治疗中应用广泛。体外研究显示几乎所有急性髓系白血病细胞上均有巨噬细胞集落刺激因子受体的表达,G-CSF不仅可以促使G0期白血病细胞进入增殖周期,使S期细胞数相对增加,有利于Ara-C的杀伤作用,还可以促使肿瘤细胞摄取更多的Ara-CTP,从而使更多的阿糖胞苷与细胞DNA结合,增加阿糖胞苷和蒽环类药物对肿瘤细胞的杀伤。联合应用去甲基化药物可增强白血病细胞对阿糖胞苷的敏感性,激活TRAIL通路,诱导急性髓系白血病细胞凋亡,进一步提高疗效。

组蛋白去乙酰化酶抑制剂(histone deacetylaseinhibitors, HDACI)作为新一代靶向抗肿瘤药物,在血液系统肿瘤及其他肿瘤中均显示出了一定疗效<sup>[28]</sup>。HDACI可抑制肿瘤细胞内高表达的HDAC活性,上调组蛋白的乙酰化水平,调控相关基因的转录,从而诱导肿瘤细胞分化或凋亡<sup>[29]</sup>。HDACi在临床应用及体外实验中均显示有抗白血病作用,联合其他化疗药物可提高治疗效果<sup>[30,31]</sup>。基础研究显示急性髓系白血病细胞存在表观遗传调控异常,HDAC与DNA甲基化相互作用,共同导致基因沉默,HDACI重新激活被DNA甲基化沉默的基因。临床前研究结果显示去甲基化药物和HDACI具有协同抗白血病作用。国外有多项去甲基化药物联合HDACI双表观调控治疗AML的临床研究,现有数据表明两者联合具有良好的疗效及耐受性。

西达本胺(chidamide)是我国自主研发的新一代酰胺类HDACI,在国内已经广泛用于治疗外周T细胞淋巴瘤,并显示出良好的疗效<sup>[32]</sup>。西达本胺主要通过抑制相关HDAC亚型以增加染色质组蛋白的乙酰化水平来引发染色质重塑,并由此改变多条信号传导通路基因表达,进而抑制肿瘤细胞周期、诱导肿瘤细胞凋亡,同时对机体细胞免疫具有整体调节活性,诱导和增强自然杀伤细胞(NK)和抗原特异性细胞毒T细胞(CTL)介导的肿瘤杀伤作用<sup>[33,34]</sup>。另外,西达本胺还可以诱导肿瘤干细胞分化、逆转肿瘤细胞的上皮间充质表型转化等,进而恢复耐药肿瘤细胞对药物的敏感性以及抑制肿瘤转移、复发等<sup>[35]</sup>。申请人既往进行的单中心西达本胺联合DCAG方案治疗复发难治急性髓系白血病的1/2期临床研究,共纳入93例患者,其中24例患者达到CR,19例患者达到CRi,总反应率46.2%,这部分患者总生存时间明显延长<sup>[19]</sup>。

#### (3) 白血病的靶向治疗

B细胞淋巴瘤因子2(B-cell lymphoma-2,BCL-2)家族是细胞内源性凋亡信号转导通路中的关键凋亡因子,维奈克拉(Venetoclax)是第一个上市的 BCL-2选择性抑制剂,目前已被批准用于老年或不能耐受强化疗的急性髓系白血病的治疗。维奈克拉单药治疗复发/难治急性髓系白血病研究中,CR/CRi率仅为19%且中位PFS很短<sup>[36]</sup>。维奈克拉并不能精确打击肿瘤细胞,而是通过凋亡机制增强抗肿瘤作用,因此,在急性髓系白血病中,维奈克拉联合其他药物至关重要。目前的研究证实,维奈克拉联合低剂量阿糖胞苷、阿扎胞苷或地西他滨可明显延长AML患者总生存时间和无事件生存时间。

从药物的组合来看,CACAG方案,包含了西达本胺、阿克拉霉素及阿扎胞苷,三者均具有表观遗传调控功能,与维奈克拉联合使用,或许不同于经典DA(柔红霉素和阿糖胞苷)方案的适用人群,可以改善初治急性髓系白血病患者对经典方案的耐药。

国内外有多项去甲基化+HDACI双表观调控治疗AML的临床研究,现有数据表明两者联合具有良好的疗效及耐受性。那么包含双表观调控治疗联合化疗的维奈克拉联合CACAG方案(阿扎胞苷+西达本胺+CAG)在急性髓系白血病的疗效值得我们进一步研究。我们拟在成人急性髓系白血病患者中进行维奈克拉联合CACAG方案和标准"3+7"方案的疗效对比研究,并通过ATAC-seq、ChIP-seq、RNA-seq多组学联合分析不同方案引起的组蛋白释放差异及其对基因表达的影响,探究AML细胞组蛋白释放状态与下游基因表达谱的特征,从而探索新的AML诱导化疗方案,改善患者预后,延长患者生存期。

#### 参考文献

- [1] YATES J, GLIDEWELL O, WIERNIK P, 等. Cytosine arabinoside with daunorubicin or adriamycin for therapy of acute myelocytic leukemia: a CALGB study[J]. Blood, 1982, 60(2): 454-462.
- [2] RAI K R, HOLLAND J F, GLIDEWELL O J, 等. Treatment of acute myelocytic leukemia: a study by cancer and leukemia group B[J]. Blood, 1981, 58(6): 1203-1212.
- [3] SCHLENK R F, FRECH P, WEBER D, 等. Impact of pretreatment characteristics and salvage strategy on outcome in patients with relapsed acute myeloid leukemia[J/OL]. Leukemia, 2017, 31(5): 1217-1220. DOI:10.1038/leu.2017.22.
- [4] CORTES J E, KHALED S, MARTINELLI G, 等. Quizartinib versus salvage chemotherapy in relapsed or refractory FLT3-ITD acute myeloid leukaemia (QuANTUM-R): a multicentre, randomised, controlled, open-label, phase 3 trial[J/OL]. The Lancet. Oncology, 2019, 20(7): 984-997. DOI:10.1016/S1470-2045(19)30150-0.
- [5] PATEL J P, GÖNEN M, FIGUEROA M E, 等. Prognostic relevance of integrated genetic profiling in acute myeloid leukemia[J/OL]. The New England Journal of Medicine, 2012, 366(12): 1079-1089. DOI:10.1056/NEJMoal112304.
- [6] RITCHIE E K, FELDMAN E J, CHRISTOS P J, 等. Decitabine in patients with newly diagnosed and relapsed acute myeloid leukemia [J/OL]. Leukemia & Lymphoma, 2013, 54(9): 2003-2007. DOI:10.3109/10428194.2012.762093.
- [7] PHILLIPS C L, DAVIES S M, MCMASTERS R, 等. Low dose decitabine in very high risk

- relapsed or refractory acute myeloid leukaemia in children and young adults [J/OL]. British Journal of Haematology, 2013, 161(3): 406-410. DOI:10.1111/bjh.12268.
- [8] 地西他滨联合改良 CAG 方案...治急性髓系白血病的临床研究\_靖彧.pdf[Z].
- [9] CHENG-YING Z, SHI-YAN L, JIAN-HUA N, 等. Clinical Resarch of Decitabine Combined with Modified CAG Regimen for Treatment of Relapsed or Refractory Acute Myeloid Leukemia[J].
- [10] DÖHNER H, ESTEY E, GRIMWADE D, 等. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel[J/OL]. Blood, 2017, 129(4): 424-447. DOI:10.1182/blood-2016-08-733196.
- [11] TEWEY K M, ROWE T C, YANG L, 等. Adriamycin-induced DNA damage mediated by mammalian DNA topoisomerase II[J/OL]. Science (New York, N.Y.), 1984, 226(4673): 466-468. DOI:10.1126/science.6093249.
- [12] NITISS J L. Targeting DNA topoisomerase II in cancer chemotherapy[J/OL]. Nature Reviews. Cancer, 2009, 9(5): 338-350. DOI:10.1038/nrc2607.
- [13] NITISS J L. DNA topoisomerase II and its growing repertoire of biological functions[J/OL]. Nature Reviews. Cancer, 2009, 9(5): 327-337. DOI:10.1038/nrc2608.
- [14] DOU L, XU Q, WANG M, 等. Clinical efficacy of decitabine in combination with standard-dose cytarabine, aclarubicin hydrochloride, and granulocyte colony-stimulating factor in the treatment of young patients with newly diagnosed acute myeloid leukemia[J/OL]. OncoTargets and Therapy, 2019, 12: 5013-5023. DOI:10.2147/OTT.S200005.
- [15] PANG B, DE JONG J, QIAO X,  $\clubsuit$ . Chemical profiling of the genome with anti-cancer drugs defines target specificities [J/OL]. Nature Chemical Biology, 2015, 11(7): 472-480. DOI:10.1038/nchembio.1811.
- [16] WIJDEVEN R H, PANG B, VAN DER ZANDEN S Y, 等. Genome-Wide Identification and Characterization of Novel Factors Conferring Resistance to Topoisomerase II Poisons in Cancer[J/OL]. Cancer Research, 2015, 75(19): 4176-4187. DOI:10.1158/0008-5472.CAN-15-0380.
- [17] PANG B, SNYDER M P. Systematic identification of silencers in human cells[J/OL]. Nature Genetics, 2020, 52(3): 254-263. DOI:10.1038/s41588-020-0578-5.
- [18] PANG B, QIAO X, JANSSEN L, 等. Drug-induced histone eviction from open chromatin contributes to the chemotherapeutic effects of doxorubicin[J/OL]. Nature Communications, 2013, 4: 1908. DOI:10.1038/ncomms2921.
- [19] WANG L, LUO J, CHEN G, 等. Chidamide, decitabine, cytarabine, aclarubicin, and granulocyte colony-stimulating factor (CDCAG) in patients with relapsed/refractory acute myeloid leukemia: a single-arm, phase 1/2 study[J/OL]. Clinical Epigenetics, 2020, 12(1): 132. DOI:10.1186/s13148-020-00923-4.
- [20] QIAO X, VAN DER ZANDEN S Y, WANDER D P A, 等. Uncoupling DNA damage from chromatin damage to detoxify doxorubicin[J/OL]. Proceedings of the National Academy of Sciences of the United States of America, 2020, 117(26): 15182-15192. DOI:10.1073/pnas.1922072117.
- [21] WOUTERS B J, DELWEL R. Epigenetics and approaches to targeted epigenetic therapy in acute myeloid leukemia[J/OL]. Blood, 2016, 127(1): 42-52. DOI:10.1182/blood-2015-07-604512.
- [22] WANG H, LIU Y C, ZHU C Y, 等. Chidamide increases the sensitivity of refractory or relapsed acute myeloid leukemia cells to anthracyclines via regulation of the HDAC3 -AKT-P21-CDK2 signaling pathway[J/OL]. Journal of experimental & clinical cancer research: CR, 2020, 39(1): 278. D0I:10.1186/s13046-020-01792-8.
- [23] OMIDBAKHSHFARD M A, WINCK F V, ARVIDSSON S, 等. A step-by-step protocol for formaldehyde-assisted isolation of regulatory elements from Arabidopsis thaliana[J/OL]. Journal of Integrative Plant Biology, 2014, 56(6): 527-538. DOI:10.1111/jipb.12151.
- [24] SHORT N J, KONOPLEVA M, KADIA T M, 等. Advances in the Treatment of Acute Myeloid Leukemia: New Drugs and New Challenges[J/OL]. Cancer Discovery, 2020, 10(4): 506-525. DOI:10.1158/2159-8290.CD-19-1011.
- [25] TORNÉ J, RAY-GALLET D, BOYARCHUK E, 等. Two HIRA-dependent pathways mediate H3.3 de novo deposition and recycling during transcription[J/OL]. Nature Structural & Molecular Biology, 2020, 27(11): 1057-1068. DOI:10.1038/s41594-020-0492-7.
- [26] WEI Y, XIONG X, LI X, 等. Low-dose decitabine plus venetoclax is safe and effective as post-transplant maintenance therapy for high-risk acute myeloid leukemia and myelodysplastic syndrome[J/OL]. Cancer Science, 2021, 112(9): 3636-3644. DOI:10.1111/cas.15048.
- [27] RITCHIE E K, FELDMAN E J, CHRISTOS P J, 等. Decitabine in patients with newly diagnosed and relapsed acute myeloid leukemia[J/OL]. Leukemia & Lymphoma, 2013, 54(9): 2003-2007. DOI:10.3109/10428194.2012.762093.
- [28] JOHNSTONE R W. Histone-deacetylase inhibitors: novel drugs for the treatment of cancer[J/OL]. Nature Reviews. Drug Discovery, 2002, 1(4): 287-299. DOI:10.1038/nrd772.
- [29] PEART M J, TAINTON K M, RUEFLI A A, 等. Novel mechanisms of apoptosis induced by histone deacetylase inhibitors[J]. Cancer Research, 2003, 63(15): 4460-4471.

- [30] FISKUS W, WANG Y, SREEKUMAR A, 等. Combined epigenetic therapy with the histone methyltransferase EZH2 inhibitor 3-deazaneplanocin A and the histone deacetylase inhibitor panobinostat against human AML cells[J/OL]. Blood, 2009, 114(13): 2733-2743. DOI:10.1182/blood-2009-03-213496.
- [31] QUINTÁS-CARDAMA A, SANTOS F P S, GARCIA-MANERO G. Histone deacetylase inhibitors for the treatment of myelodysplastic syndrome and acute myeloid leukemia[J/OL]. Leukemia, 2011, 25(2): 226-235. DOI:10.1038/leu.2010.276.
- [32] 《中国肿瘤临床》文章荐读:... 国专家共识(2018 年版)\_本刊编辑部. pdf[Z].
- [33] NING Z Q, LI Z B, NEWMAN M J,  $\stackrel{\text{cond}}{\Rightarrow}$ . Chidamide (CS055/HBI-8000): a new histone deacetylase inhibitor of the benzamide class with antitumor activity and the ability to enhance immune cell-mediated tumor cell cytotoxicity[J/OL]. Cancer Chemotherapy and Pharmacology, 2012, 69(4): 901-909. DOI:10.1007/s00280-011-1766-x.
- [34] YAO Y, ZHOU J, WANG L, 等. Increased PRAME-specific CTL killing of acute myeloid leukemia cells by either a novel histone deacetylase inhibitor chidamide alone or combined treatment with decitabine[J/OL]. PloS One, 2013, 8(8): e70522. DOI:10.1371/journal.pone.0070522. [35] ZHOU Y, PAN D S, SHAN S, 等. Non-toxic dose chidamide synergistically enhances platinum-induced DNA damage responses and apoptosis in Non-Small-Cell lung cancer cells[J/OL]. Biomedicine & Pharmacotherapy = Biomedecine & Pharmacotherapie, 2014, 68(4): 483-491. DOI:10.1016/j.biopha.2014.03.011.
- [36] KONOPLEVA M, POLLYEA D A, POTLURI J, 等. Efficacy and Biological Correlates of Response in a Phase II Study of Venetoclax Monotherapy in Patients with Acute Myelogenous Leukemia[J/OL]. Cancer Discovery, 2016, 6(10): 1106-1117. DOI:10.1158/2159-8290.CD-16-0313.

#### 二、 研究目的及意义

#### ①研究目的: 提升急性髓系白血病患者诱导化疗方案疗效, 改善患者预后

急性髓系白血病(acute myeloid leukemia,AML)是成人最常见的急性白血病类型,含蒽环类药物(例如柔红霉素和去甲氧柔红霉素)的传统"3+7"方案是治疗急性髓系白血病最重要最常用的诱导方案之一。该方案可使60%-70%的初治白血病患者获得血液学缓解,但30%-40%的初治患者对于传统蒽环类方案原发耐药,治疗效果极差。而且,获得缓解的患者中,30%-40%患者后期也会出现药物耐药,导致白血病复发。难治或复发耐药急性髓系白血病患者生存率极低,是白血病治疗中最棘手的问题之一,亟须寻找新的诱导化疗方案改善AML患者预后。

#### <u>②研究意义:</u>

传统"3+7"的AML诱导化疗方案为阿糖胞苷联合不同的蒽环类药物如柔红霉素或去甲氧柔红霉素,是NCCN(National Comprehensive Cancer Network,美国国立综合癌症网络)等各大指南的一线推荐。蒽环类药物包括阿霉素(adriam ycin)、柔红霉素(daunorubicin)、去甲氧柔红霉素(idarubicin)和阿克拉霉素(aclarubicin)等(Figure 1),其分子结构中存在一个相同的苷元环,机制是通过抑制拓扑异构酶II(topoisomerase II,Topo II),影响DNA拓扑结

构转换,从而阻碍复制、转录和DNA修复,或者嵌入DNA双链碱基之间形成稳定复合物抑制DNA复制和RNA合成。

Figure 1 临床常用蒽环类药物的化学结构;

20世纪70年代起,DA或IA方案(3+7方案)成为了AML的标准诱导治疗方案,在年轻成人AML患者中完全缓解率达到60-70%。近40年研究中发现通过增强化疗药物剂量、增加化疗药物种类或联合其他靶向药物,可以提高部分携带特定分子学异常的AML患者的治疗反应率,但成人AML总体预后并无明显改善。且AML多种化疗药物耐药的机制存在共同性,如蒽环类药物、嘧啶类抗代谢药物阿糖胞苷等存在共同的耐药机制。而且白血病细胞一旦对一种药物产生耐药,往往多种药物皆存在耐药情况。

AML的治疗决策在近几十年主要围绕着化疗方案的强度和不同化疗药物的组合,缺少突破性进展。虽然国内外不断有治疗AML的新药上市,包括靶向BCL-2(B-cell lymphoma-2,B淋巴细胞瘤-2)的维奈克拉,靶向FLT3(Fms-like tyrosine kinase, FMS样的酪氨酸激酶3)的米哚妥林和吉瑞替尼,靶向IDH1(i socitrate dehydrogenase soluble 1,可溶性异柠檬酸脱氢酶1)、IDH2的艾伏尼布和恩西地平,针对CD33的GO以及柔红霉素和阿糖胞苷的脂质体复合物CPX-351及IDH2抑制剂等。新药在临床取得了一定的效果,改善了部分携带特定分子学异常、老年患者及不能耐受强化疗患者的治疗效果,但均替代不了蒽环类药物

的重要地位,且初诊的成人AML患者总体预后并无明显改善,仍有约30%的患者因诱导失败或疾病复发而成为复发难治急性白血病。

因此,克服原发或复发后的耐药,寻找新的治疗方案提高急性髓系白血病患者诱导化疗的缓解率、提高该类患者治疗疗效、改善患者预后生存有重大的研究价值。

#### 三、 研究内容

#### (1) 开展前瞻性随机对照临床试验

收入初治AML患者160例,前瞻随机入组,应用经典"3+7"的IA方案(去甲氧柔红霉素+阿糖胞苷)或CACAG+维奈克拉方案(西达本胺+阿扎胞苷+阿克拉霉素+阿糖胞苷+粒细胞集落刺激因子+维奈克拉),比较两组的疗效和安全性。治疗方案如下:

患者签署知情同意后进入随机化程序,随机分为试验组和对照组。

**对照组**:接受经典IA治疗方案,整个试验治疗期共1周,每4周是一个治疗周期,总共2个疗程。

- ①去甲氧柔红霉素 (Idarubicin): 8-10mg/m2 第1至3天应用;
- ②阿糖胞苷 (Ara-C): 100mg/m2 q12h第1至7天应用。

试验组:接受CACAG+维奈克拉治疗方案,整个试验治疗期共1周,每4周是一个治疗周期,总共2个疗程。

- ①西达苯胺(Chidamide): 30 mg, 每周两次, 总共应用2次;
- ②阿扎胞苷(Azacitidine): 75 mg/m2 第1至7天应用;
- ③阿糖胞苷 (Ara-C): 75-100 mg/m2 q12h第1至7天应用;
  - ④阿柔比星(Aclarubicin): 20 mg/m2, 第1, 第3, 第5天应用;
- ⑤重组人粒细胞集落刺激因子(G-CSF): 300ug/天,直至中性粒细胞恢复,白细胞≥20000/ul停用。
- ⑥维奈克拉(Venetoclax): 100mg 第1天, 200mg 第2天, 400mg 第3-14天, 与唑类药物联用, 减量为100mg/天;

本试验的治疗周期是 2 周期 (8 周),如第1疗程治疗后评估未达到PR,则退出实验组,根据指南给予更换其他治疗方案。

前瞻随机对照研究试验流程图如下:



#### (2) 通过多组学分析探索诱导治疗方案的表观遗传学调控新机制

- ①采用ATAC-seq、ChIP-seq、RNA-seq多组学技术,展示不同药物治疗方案下AML患者的组蛋白释放谱及修饰谱的用药前后差异。
- ②通过ATAC-seq、ChIP-seq、RNA-seq多组学联合分析不同药物引起的组蛋白释放对基因表达的影响,通过信号通路富集分析揭示不同治疗方案引起组蛋白释放引起的差异信号通路。
- ③多组学联合分析诱导化疗耐药患者 AML 细胞组蛋白释放状态与下游基因表达谱的特征。

#### 四、研究设计

- (1) CACAG+维奈克拉方案治疗初诊急性髓系白血病的前瞻性、随机对照临床研究
  - ① 研究类型及分组: 开放性、前瞻性、随机对照研究。

试验组: 80例

对照组:80例

- ② 试验对象:严格按照前述的入组标准和排除标准选择初治AML患者进入临床试验。
  - ③ 治疗方案:

对照组:接受经典"3+7" IA诱导缓解方案

IA方案整个试验治疗期共1周,每4周是一个治疗周期,总共2个疗程。

去甲氧柔红霉素 (Idarubicin): 8-10mg/m2 第1至3天应用;

阿糖胞苷 (Ara-C): 100mg/m2 q12h第1至7天应用。

试验组:接受CACAG+维奈克拉诱导缓解方案

CACAG+维奈克拉方案整个试验治疗期共1周,每4周是一个治疗周期,总共1个疗程。

- ①西达苯胺(Chidamide): 30 mg,每周两次,总共应用2次;
- ②阿扎胞苷(Azacitidine): 75 mg/m2 第1至7天应用;
- ③阿糖胞苷 (Ara-C): 75-100 mg/m2 q12h第1至7天应用;
- ④阿柔比星(Aclarubicin): 20 mg/m2, 第1, 第3, 第5天应用;
- ⑤重组人粒细胞集落刺激因子(G-CSF): 300ug/天,直至中性粒细胞恢复,白细胞≥20000/u1停用;
- ⑥维奈克拉 (Venetoclax): 100mg 第1天, 200mg 第2天, 400mg 第3-14 天, 与唑类药物联用, 减量为100mg/天;

本试验的治疗周期是 2 周期(8 周),如第1疗程治疗后评估未达到PR,则退出实验组,根据指南给予更换其他治疗方案。

(2) 药物诱导组蛋白释放后,新填充组蛋白的表观遗传修饰特征研究

- ①收取初治AML病人用药前后骨髓标本,用聚蔗糖一泛影葡胺(Ficoll-1sopaque)淋巴细胞分离液梯度离心提取病人单个核细胞,采用磁珠分选CD33+白血病细胞进行体外培养,用去甲氧柔红霉素、阿克拉霉素、依托泊苷、柔红霉素处理K562、HL60和提取的原代细胞4h后用DMS0、FBS彻底清洗药物后继续于RPMI 1640培养基培养,留取用药4h、撤药后0h、4h、8h、24h时间节点样本进行后续实验,并设置空白对照。
- ②荧光蛋白标记组蛋白:构建光激活绿色荧光蛋白(photo-activatable green fluorescent protein)慢病毒载体,药物处理前转染细胞,在N端标记组蛋白H2A、H2B和H2AX,在C端用PAGFP标记H3和H4,用G418进行富集筛选稳定表达修饰后组蛋白的细胞株。
- ③激光扫描共聚焦显微镜(confocal laser scanning microscope, CLSM)观察组蛋白动向。每个时间节点样本用激光扫描共聚焦显微镜观察60min并记录 0min、15min、30min、60min组蛋白释放情况。
- ④FAIRE-seq和ATAC-seq检测染色质可及性。用FAIRE-seq和ATAC-seq 检测不同药物处理和不同时间节点的染色质可及性变化,揭示药物引起的组蛋白释放。
- ⑤ChIP-seq检测用药前后组蛋白表观遗传特征的变化。采用ChIP-seq方法 检测用药前后各时间点组蛋白修饰特征的变化,通过用药前后ChIP-seq变化找出 用药后组蛋白修饰的变化和撤药后组蛋白修饰的变化,相关检测位点如下表:

| Histone H3 | Histone H3.3 | Histone H2A.Z | Histone H3K4me3 |
|---|---|---|---|
| Histone H3K4me2 | Histone H3K4me1 | Histone H3K9me3 | Histone H3K9me2 |
| Histone H3K9me1 | Histone<br>H3K27me3 | Histone<br>H3K27me2 | Histone H3K27me1 |
| Histone<br>H3K36me3 | Histone<br>H3K27me2 | Histone<br>H3K27me1 | Histone H3K79me2 |
| Histone H3K14ac | Histone H3K18ac | Histone H3K27ac | Histone H3K9ac |
| Histone H3K36ac | Histone H4K12ac | Histone H2BK5ac | Histone<br>H2BK120ac |

| Histone H3K56ac | Histone |
|-----------------|------------|
| | H2AK119ub1 |

⑥将ATAC-seq、FAIRE-seq、ChIP-seq和共聚焦激光扫描显微镜联合分析,观察蒽环类药物引起组蛋白释放及其引起的组蛋白修饰的变化,观察撤药后新填补组蛋白引起的组蛋白修饰的变化。通过机器学习将表观遗传状态与临床疗效关联分析。

# (3) 化疗药物诱导组蛋白释放后,下游基因表达谱的变化特征及与组蛋白表观 遗传修饰特征的融合分析

- ①RNA-seq检测组蛋白释放后对基因表达的影响。对用药前后K562、HL60、AML原代细胞进行RNA-seq分析药物引起的基因表达的变化。
- ②联合ATAC-seq、FAIRE-seq、ChIP-seq和RNA-seq数据,找到药物处理后差异表达基因所在染色质全长区域的组蛋白释放的变化,筛选出组蛋白释放引起的差异表达基因,通过ChIP-seq分析差异基因组蛋白释放区域内有哪些组蛋白修饰在用药前后存在差异,因而找到调控组蛋白释放进而调控基因表达的表观遗传修饰的特征性修饰。
- ③对差异基因进行通路富集分析,找到用药后引起的通路表达的变化。这些差异基因和通路是研究不同治疗方案疗效差别的重要位点,通过联合分析可以将的研究范围极大地缩小,更进准的找到引起耐药的差异通路和治疗的靶点。
- ④进行RNA-seq、ATAC-seq分析原代急性髓系白血病细胞组蛋白释放状态与下游基因表达谱的特征。通过ATAC-seq(scATAC-seq)对不同细胞系和不同时间节点的标本进行分析,对蒽环类药物引起的组蛋白释放的细胞类型和状态进行鉴定和聚类,分析出所有差异表达活跃转录的调控序列。发现具有细胞特异性活性的细胞特异性结合位点和差异表达基因及通路,通过motif富集分析找到特异性转录调节因子。将表观遗传状态与临床疗效关联分析。

#### (4) 观察指标:

- ①主要疗效指标: 1疗程复合完全缓解率 (complete remission, CRc);
- ②次要疗效指标: 1疗程完全缓解伴血细胞不完全恢复率(CRi),1疗程部分缓解率(PR),1疗程总反应率(ORR),1疗程完全缓解率(CR)、2疗程完全缓解性血细胞不完全恢复率(CRi),2疗程部分缓解率(PR)、微小病变残留(

- MRD)、2疗程无事件生存期(EFS)、总生存时间(OS);
- ③安全性指标:不良事件:类型、发生率、与试验药物的关系、严重程度; 实验室检查异常:临床实验室检查的异常类型、发生率、与试验药物的关系、严 重程度; 3~4 级临床不良事件和实验室检查异常的发生率。
  - ④疗效评价间隔:每个疗程治疗结束14-21天进行评价;
  - ⑤疗效评价手段: 外周血及骨髓形态学、基因定量检测、白血病免疫分型;
  - ⑥疗效评价标准:

| 完全缓解 (CR) | 临床无白血病细胞浸润所致的症状和体征 |
|-----------|-------------------------------|
| | ; 血象: Hb≥ 100g/L (男) 或≥ 90g/L |
| | (女及儿童),中性粒细胞绝对值≧ 1.5 |
| | × 109/L, 血小板≥ 100× 109/L。外周 |
| | 血白细胞分类中无白血病细胞;骨髓象: |
| | 原粒细胞 I 型+II 型(原始单核+幼稚单 |
| | 核细胞)≦ 5%,红细胞及巨核系正常; |
| CRi | 骨髓中原始细胞<5%,不依赖输血,但持 |
| | 续性血细胞不恢复; |
| 部分缓解 (PR) | 骨髓中原始细胞减少大于 50%以上,且比 |
| | 例达到 5%-25%,且外周血细胞计数恢复 |
| | 正常; |
| ORR | CR+PR |
| 复发 | 完全缓解(CR)后外周血再次出现白血病 |
| | 细胞或骨髓中原始细胞5%(除外巩固化疗 |
| | 后骨髓再生等其他原因)或髓外出现白血 |
| | 病细胞浸润; |
| PFS | 从试验治疗开始到第一次出现疾病进展的 |
| | 时间长度; |
| OS | 从试验治疗开始到死亡或随访结束的时间 |
| | 长度; |
| 安全性分析 | 详细描述发生血液或非血液毒性反应的病 |
| | 例情况,计算不同事件的发生率,计算各 |
| | 事件严重程度的构成比。 |
| | 1 |

#### (5) 随访计划

在最后一例病人入组完成治疗,并随访3个月后作为数据的截尾日。所有病例 将继续随访并观察记录远期疗效。所有患者在试验期需进行的评估内容及时间, 请参见下页的随访时间内容表:

#### 试验流程表

| 试验阶段 | 筛选期 | 治疗周期 | | 试验结束访视 <sup>8</sup> | 生存随访 <sup>9</sup> |
|---|---|---|---|---|---|
| 治疗疗程 | | 1 | 2 | | |
| 随访次数 | 1 | 2 | 3 | 5 | |
| 周/天 | D-7至DO | D1-D28 | D29-D58 | 试验结束后2<br>周内 | 每2-3月1次<br>直至试验结<br>束 |
| 签署知情同意书1 | × | | | | |
| 核查入选/排除标准 | × | | | | |
| 人口统计学资料 | × | | | | |
| 病史/手术史 | × | | | | |
| 体格检查 | × | × | × | × | |
| 生命体征 | × | × | × | × | |
| ECOG体力状态 | × | × | × | × | |
| 输血记录 | × | 根据病情随时记录 | | | |
| 体温记录 | × | 根据病情随时记录 | | | |
| 血常规 | ×2 | 每周至少3次,根据病<br>情需要增加 | | × | |
| 血生化(肝肾<br>功、空腹血糖、<br>电解质) | ×2 | 每周至少3次根据病情<br>需要增加 | | | |
| 血清病原学检测 | × | | 命血情况随时<br>金测 | | |
| 凝血功能³ | × | × | × | | |

| 淋巴细胞亚群<br>及细胞因子、<br>GVHD情况 | × | × | × | | |
|----------------------------|---|-----|---|---|---|
| 12导联心电图 | × | 必要时 | | | |
| 尿常规 | × | × | × | | |
| 心脏超声 | × | 必要时 | | | |
| 肿瘤评估 4 | × | × | × | × | × |
| 妊娠试验 5 | × | | | | |
| 基因检测样本。 | × | | | | |
| 记录更换治疗方式 | | | | × | |
| 发放药物 | | × | × | | |
| 回收药物 | | | | | |
| 记录不良事件 | | | | × | |
| 记录合并用药 | × | | | × | |
| 生存期及后续<br>疾病治疗情况 | | | | | × |

#### 注:

- 1. 知情同意书必须在进入筛选期前获得。
- 2. 筛选期的血常规、血生化检查需在接受试验治疗前 1 周内进行。
- 3. 每4 周至少检查1 次,可根据病情需要增加频率。
- 4. 包括骨髓细胞形态学分析、免疫分析等。
- 5. 适用于育龄期女性。
- 6. 在初诊时采集 5ml 骨髓样本,提取单个核细胞, -80 摄氏度冰箱保存;
- 7. 每个访视周期的窗口期为±2天。若患者治疗过程中有暂停用药,新周期开始的定义是服用新周期的试验药物。 C: 周期; W: 周; D: 天。
- 8. 结束试验治疗后2周内,需要返院进行结束治疗的访视。
- 9. 可以通过电话随访完成

总生存期 (OS) 为次要疗效指标,为获得 OS 数据,还应该对试验结束后的患者进行生存随访,每2-3 个月电话或当面随访患者的生存情况,并将结果记录在 CRF 的试验完成后随访页。

#### (6) 统计分析方法

采用电子病例报告表(EDC),由研究者或者研究者指定人员参照原始资料如实录入。详细描述发生血液或非血液毒性反应的病例情况,计算不同事件的发生率,计算各事件严重程度的构成比,进行安全性分析。所有统计分析采用SAS 9.2 完成,计量数据采用均数、标准差、中位数、最大值、最小值描述,计数数据采用频数、百分比描述。主要疗效指标一疗程完全缓解(CR)率进行卡方等检验。次要疗效指标1疗程完全缓解伴血细胞不完全恢复率(CRi)、1疗程部分缓解率(PR)、1疗程总反应率(ORR)、2疗程完全缓解率(CR)、2疗程完全缓解伴血细胞不完全恢复率(CRi)、2疗程完全缓解伴血细胞不完全恢复率(CRi)、2疗程完全缓解伴血细胞不完全恢复率(CRi)、2疗程完全缓解体血细胞不完全恢复率(CRi)、2疗程的份缓解率(PR)、微小病变残留(MRD)、2疗程无事件生存期(EFS)、总生存时间(OS)进行卡方等检验,计算 95%CI。 采用Kaplan-Meier 法估计总生存时间(OS)在各时间点上的生存率、中位生存时间及其 95%CI,并绘制生存曲线图。

#### (7) 数据采集和管理

研究者必须妥善处理所有临床试验过程中获得的数据,以保证参与临床试验的患者的权利和隐私。研究者必须同意监查员/稽查员/视察员对所需要的临床试验资料进行查阅和审核,以便验证原始资料的准确性和了解试验的进展情况。如果不能对原始记录进行验证,则研究者应同意协助监查员/稽查员/视察员对数据的质量进行进一步的确认。考虑到门诊治疗随访的患者,除患者入组信息,肿瘤评估,给药记录,不良事件和实验室检查等信息需在门诊病历记录外, CRF 记录的部分信息如生命体征将作为原始数据保存。试验资料将按照 GCP 要求妥善保管在各试验中心,包括能对受试者身份进行确认的文件(如原始的有签名的知情同意书、原始医疗记录)、试验用药物发放/回收记录等。所有试验文件应保存至本临床试验结束后 5 年。

#### 五、 试验流程图(技术路线图)

# 初治成人急性髓系白血病患者中标准 "3+7" 方案与维奈克拉联合CACAG方案的多中心前瞻随机对照研究



六、 试验对象入选/排除标准、退出/中止标准

#### 1. 纳入标准:

- ①自愿参加临床研究;本人或法定监护人完全了解、知情本研究并签署知情同意书(ICF);愿意遵循并能完成所有试验程序;
  - ②筛选时年龄14-75岁,性别不限:
  - ③患者为初治 AML,诊断符合2021年版中华医学会标准;
  - ④无严重过敏体质;
  - ⑤肝功能: ALT和AST≤2.5倍正常值高限, 胆红素≤2倍正常值高限:
  - ⑥肾功能: 肌酐≤正常值高限; 没有难以控制的感染及严重精神心理疾患;
  - ⑦体力评分为0-3(ECOG),预计生存期大于等于 4 个月。

#### 2. 排除标准:

- ①存在对受试药物过敏及禁忌症的患者:
- ②妊娠期、哺乳女性患者;
- ③有活动性感染;
- ④吸烟长期酗酒以致影响试验结果评价的患者;
- ⑤患者精神疾或其他病情无法获得知情同意,不能配合完成治疗和检查步骤的要求;
  - ⑥机体重要器官外科手术后未满 6 周者;
- ⑦肝功能异常,总胆红素>正常上限的 1.5 倍, ALT/AST>正常值上限 2.5 倍或肝受侵患者 ALT/AST>正常值上限 5 倍;肾功能异常,血肌酐>正常值上限 1.5 倍;

⑧研究者认为不适合本次临床试验(如依从性差、药物滥用等)。

#### 七、 常见不良反应/严重不良反应的处理预案

#### 1. 常见不良反应处理预案

任何药物均有不良反应。根据前期临床研究资料,本实验药物常见的不良反应 为消化道反应(厌食、恶心、腹泻、呕吐和胃肠胀气等)、骨髓抑制(血小板降低、 白细胞或中性粒细胞降低、血红蛋白降低)、乏力。如受试者出现骨髓抑制,则研 究者应根据血象变化情况,及时给予粒细胞集落刺激因子,刺激中性粒细胞恢复, 必要时输入红细胞悬液或血小板,改善贫血症状,预防出血,同时加强环境保护, 预防各种感染。如受试者出现过敏反应,则受试者根据患者临床表现,首先及时停 药,并给予抗过敏药物,必要时加用糖皮质激素,如出现严重过敏应,及时加用生 命体征监护,积极加强液体支持,并给予改善微循环,维持血压等治疗。如出现肝 肾功能损伤, 予积极保肝、水化、碱化,密切监测肝肾功能变化。如受试者出现 胃肠道反应,则予止吐、抑酸、保护胃黏膜、止泻等对症治疗。

#### 2. 严重不良反应处理预案

临床试验过程中发生符合下列情况中的一种或以上事件时,可判定为

- ① 严重不良事件 (Serious Adverse Event, SAE) 致死;
- ② 危及生命:
- ③ 非社会因素(如保险报销)导致的住院治疗或延长住院时间的医学事件;
- ④ 导致持续的或严重残疾/功能障碍;
- ⑤ 受试者的后代出现先天性异常/出生缺陷:
- ⑥ 重大医学事件;
- ⑦ 所有妊娠事件均参照严重不良事件报告。

在临床试验过程中如发生严重不良事件,研究者应立即对受试者采取适当的 救治措施并记录于原始资料中,于 24 小时内报告试验中心主要研究者及伦理委 员会和申办者。研究者须认真逐项填写严重不良事件报告表, 并在报告上签名及 注明日期。

#### 八、 数据统计方法

采用电子病例报告表(EDC),由研究者或者研究者指定人员参照原始资料如实录入。详细描述发生血液或非血液毒性反应的病例情况,计算不同事件的发生率,

计算各事件严重程度的构成比,进行安全性分析。所有统计分析采用 SAS 9.2 完成,计量数据采用均数、标准差、中位数、最大值、最小值描述,计数数据采用频数、百分比描述。主要疗效指标一疗程完全缓解(CR)率进行卡方等检验。次要疗效指标1疗程完全缓解伴血细胞不完全恢复率(CRi)、1疗程部分缓解率(PR)、1疗程总反应率(ORR)、2疗程完全缓解率(CR)、2疗程完全缓解伴血细胞不完全恢复率(CRi)、2疗程部分缓解率(PR)、微小病变残留(MRD)、2疗程无事件生存期(EFS)、总生存时间(OS)进行卡方等检验,计算 95%CI。 采用Kaplan-Meier 法估计总生存时间(OS)在各时间点上的生存率、中位生存时间及其 95%CI,并绘制生存曲线图。

### 中国人民解放军总医院第五医学中心 伦理审查小组审查批件

地址: 北京市丰台区东大街 8 号 郎編: 100071 电话: 010-66947798 传真: 010-66947798

#### 批件号: KY-2024-3-40-2

| 项目名称 | | 台成人急性髓系白血病患者中的多中心前瞻随机对照研究 | 标准 "3+7" | 方案与维奈克 | 拉联合 CA | CAG为 |
|------|----|---------------------------|----------|----------|--------|------|
| 申办者 | | 中国人民解放军总医院<br>第五医学中心 | 研究科室 | 血液内科 | 研究者 | 窦立萍 |
| 送审资料 | 1. | 复审申请表<br>知情同意书(版本号: 1.1, | 版本日期: | 2024年4月1 | 0日) | |

审查方式: 快速审查

审查时间: 2024年4月12日

同意2人、必要的修改后同意0人、不同意0人

#### 伦理审查小组审查意见:

经伦理委员会审查认为本研究符合要求,同意开展。批件有效期为6个

组长签字: 多んし

- 1. 本院发生的 SAE/SUSAR, 研究期间安全性更新报告应及时递交本伦理审查小组
- 2. 研究过程中若变更主要研究者或对研究方案、知情同意书、招募材料等的任何能改。 经伦理审查小组审查获得批准后方可执行:
- 3. 按照初始审查批准的批件有效期及时递交年度/定期跟踪审查报告;
- 4. 发生方案违背时及时逆交不依从/违背方案报告:
- 5. 暂停或提前终止研究时应及时递交暂停或提前终止研究报告:
- 6. 完成研究后递交结题报告。